CLINICAL TRIAL: NCT00035815
Title: Insulin-like Growth Factor-1 in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Insulin-like Growth Factor-1 in Amyotrophic Lateral Sclerosis (ALS) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); ALS Association (Other); Cephalon (Industry)
Responsible Party: Eric Sorenson, M.D., Department of Neurology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1461-01; R01NS042759 (NIH)
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; ALS; progressive weakness; insulin-like growth factor-1; IGF-I; Myotrophin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Insulin-Like Peptides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGF-1 (Active Comparator): Insulin like growth factor, type 1 will be given 0.05 mg per kg body weight subcutaneously twice daily
  Interventions: Drug: Insulin like growth factor, type 1
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin like growth factor, type 1 — 0.05 mg per kg body weight given subcutaneously twice daily
  Other Names: Mycotrophin
  Arms: IGF-1
Drug: Placebo — The placebo represented the inert suspension vehicle for the IGF-1. It was given as equal volume as the active drug based upon body weight, subcutaneously twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this multicenter study is to determine if insulin-like growth factor-1 (IGF-I) slows the progressive weakness in amyotrophic lateral sclerosis (ALS) patients. Study participants will be followed for 2 years once enrolled. They will receive either placebo or the active IGF-I. Examinations will take place at approximately 6-month intervals.

DETAILED DESCRIPTION:
The objective of this trial was to determine whether IGF-1 (MyotrophinTM) slows progression of weakness in amyotrophic lateral sclerosis (ALS). Three hundred thirty patients with ALS from 20 medical centers participated in this double blind, placebo-controlled two-year study. Half the patients received IGF-1 and the other half received placebo. The drug will be administered twice a day.

ALS is a neurodegenerative disorder that causes progressive muscle weakness and loss of motor neurons. IGF-1 is a neurotrophic factor essential for normal development of the nervous system and shows protection of motor neurons in animal models and cell culture systems. It is thought to block cell death pathways and promote muscle re-innervation and axonal growth and regeneration.

ELIGIBILITY:
Inclusion Criteria

Patients entering this study:

* Are between the ages of 18-80 years old.
* Legal residents of the United States or Canada.
* Have a history of a chronic onset of a progressive motor weakness of less than 24 months duration.
* Fulfill El Escorial criteria of probable or definite ALS.
* If female, are surgically sterile, two years postmenopausal, or if of child-bearing potential, must be using a medically acceptable method of birth control and agree to continue use of this method for the duration of the study. Acceptable methods include a barrier method with spermicide, oral contraceptives (normal doses are acceptable; low dose oral contraceptives or contraceptive implants must be used with a barrier method), intrauterine device (IUD), or abstinence. Have a negative pregnancy test.
* Are able to comply with protocol requirements.
* Can provide written informed consent.
* Have a manual muscle testing score of less than 8.
* Have a forced vital capacity by pulmonary function testing *60% predicted.

Exclusion Criteria:

Patients entering this study will not:

* Have any of the following conditions:renal disease (Creatine > 2.0) or other active systemic disease
* Have any clinically significant abnormalities on the prestudy laboratory evaluation, physical examination, ECG, chest x-ray or ophthalmologic exam.
* Have any clinically significant medical condition (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure) that, in the opinion of the investigator, would compromise the safety of patient.
* Have Type I or Type II diabetes.
* Have a history of cancer including melanoma with the exception of localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline) and carcinoma in-situ of the cervix (women only).
* Have used an investigational drug within 30 days of baseline visit.
* Have had a tracheostomy.
* Have a Beck's Depression Inventory score * 12.
* Have legal residency outside of the United States or Canada.
* Be pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sorenson, M.D., Principal Investigator — Department of Neurology, Mayo Clinic
Locations (20):
- United States (19):
  - Mayo Clinic in Scottsdale, Scottsdale, Arizona
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic in Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Beth Israel Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
  - Froedtert and Medical College Clinics, Milwaukee, Wisconsin
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Howe CL, Bergstrom RA, Horazdovsky BF. Subcutaneous IGF-1 is not beneficial in 2-year ALS trial. Neurology. 2009 Oct 13;73(15):1247; author reply 1247-8. doi: 10.1212/WNL.0b013e3181b26ae6. No abstract available. PMID 19822878
- [Result] Sorenson EJ, Windbank AJ, Mandrekar JN, Bamlet WR, Appel SH, Armon C, Barkhaus PE, Bosch P, Boylan K, David WS, Feldman E, Glass J, Gutmann L, Katz J, King W, Luciano CA, McCluskey LF, Nash S, Newman DS, Pascuzzi RM, Pioro E, Sams LJ, Scelsa S, Simpson EP, Subramony SH, Tiryaki E, Thornton CA. Subcutaneous IGF-1 is not beneficial in 2-year ALS trial. Neurology. 2008 Nov 25;71(22):1770-5. doi: 10.1212/01.wnl.0000335970.78664.36. PMID 19029516
- See also: The ALS Association website. — http://www.alsa.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from 20 medical centers from June 2003 to August 2005.
Pre-assignment Details: Patients were randomized and initiated on treatment at the time of enrollment.
Groups:
- IGF-1: The insulin-like growth factor type 1 (IGF-1) arm was the active treatment group. They received 0.05 mg/kg body weight administered subcutaneously twice daily.
- Placebo: Placebo group received the equal volume (based on kg of body weight) of the inert suspension vehicle in which the IGF-1 was suspended.
Period: Overall Study
Arm/Group | IGF-1 | Placebo
Started | 167 (Enrollment began June 2003, accrual was for 2 years, follow-up period was 2 years.) | 163 (Enrollment began June 2003, accrual was for 2 years, follow-up period was 2 years.)
Completed | 150 | 152
Not Completed | 17 | 11
Not completed — Withdrawal by Subject | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- IGF-1: The IGF-1 arm was the active treatment group. They received 0.05 mg/kg body weight administered subcutaneously twice daily.
- Total: Total of all reporting groups
Arm/Group | IGF-1 | Placebo | Total
Number analyzed (Participants) | 167 | 163 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 129 | 264
  >=65 years | 32 | 34 | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.2) | 54.8 (11.2) | 54.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 120
  Male | 110 | 100 | 210
Region of Enrollment [Number; unit: participants]
  United States | 167 | 163 | 330

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Composite Manual Muscle Testing (MMT) Score
Description: The primary outcome measure was the rate of change in the MMT score. MMT involved the examination of 34 muscle groups with standard positioning. The final MMT score represented an average of the 34 muscles examined, and ranged from 10 to 0(10 normal strength, 0 paralyzed). The individual muscle score was based on the medical research council (MRC) grading scale (1-5) modified to a 10 point system corresponding to the MRC modifications of plus and minus (5, 5-,4+,4,4-,3+,3, 3-,2,1,0; with 5 being normal strength and 0 paralyzed).
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: MMT units per month
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 167 | 163
MMT units per month | 0.44 (0.57) | 0.39 (0.39)
Statistical Analysis 1: Comparison: IGF-1 vs Placebo; Analysis of MMT was calculated as a ratio of change from baseline to last follow-up to time to duration until last follow-up. For the patients that died during the study period, the last follow-up time was considered as the time of death with a zero score for MMT measurement. Analysis was performed using intention to treat approach. Comparison of rate of change in MMT scores between the placebo and IGF-1 group was made using two sample t-test or Wilcoxon rank sum test as appropriate; Test type: Superiority or Other; p = 0.529, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants Alive and Tracheostomy-free at 24 Months
Description: Patients who elected to proceed to tracheostomy were assessed the month of their procedure. Subjects who continuously utilized non-invasive positive pressure ventilation for greater than 10 days were assessed as being ventilator-dependent on the first day they began continuous Non Invasive Positive Pressure Ventilation (NIPPV). All subjects were followed for the 24 month time period.
Time Frame: baseline to 24 months
Measure: Number; unit: participants
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 167 | 163
participants | 93 [0.77 to 1.4] | 90 [1 to 1]
Statistical Analysis 1: Comparison: IGF-1 vs Placebo; Patients who elected to proceed to tracheostomy were assessed on the day of their procedure. Subjects who continuously utilized NIPPV for greater than 10 days were assessed as being ventilator-dependent on the first day they began continuous NIPPV. Survival between groups was compared using the Cox-proportional Hazards model; Test type: Superiority or Other; p = 0.415, Regression, Cox; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.77 to 1.4]

3. Secondary Outcome: Rate of Change in ALS Functional Rating Scale.
Description: The final secondary outcome measure was the rate of change in the ALS Functional Rating Scale (ALSFRS-r) score. The ALSFRS-r was completed at each visit (randomization and then at 3, 6, 12, 18 and 24 months post-randomization). This is a scale from 0 to 48 assessing functional impairment in 12 clinically relevant areas in ALS. Forty-eight is normal with full function and zero is total loss of function in all clinical functions. As with the MMT scores a score of 0 was imputed on the day of death. Analysis of the ALSFRS-r scores as a secondary outcome was performed in similar manner as MMT score.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale per month
Arm/Group | IGF-1 | Placebo
Number analyzed (Participants) | 167 | 163
Units on a scale per month | 2.5 (3.2) | 2.2 (2.1)
Statistical Analysis 1: Comparison: IGF-1 vs Placebo; The final secondary outcome measure was the rate of change in the ALSFRS-r score. The ALSFRS-r was completed at each visit (randomization and then at 3, 6, 12, 18 and 24 months post-randomization). As with the MMT scores a score of 0 was imputed on the day of death. Analysis of the ALSFRS-r scores as a secondary outcome was performed in similar manner as MMT score; Test type: Superiority or Other; p = 0.321, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 years of follow-up
Arm/Group | IGF-1 | Placebo
Serious Adverse Events (participants affected / at risk) | 18/167 | 12/163
Other Adverse Events (participants affected / at risk) | 103/167 | 92/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGF-1 (N=167) | Placebo (N=163)
Thrombotic events (Vascular disorders) | 18 (18) | 12 (12) — Serious thrombotic events
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGF-1 (N=167) | Placebo (N=163)
Site reactions (Skin and subcutaneous tissue disorders) | 88 (88) | 92 (92)
Headache (Nervous system disorders) | 22 (22) | 22 (22)
Hepatotoxicity (Hepatobiliary disorders) | 14 (14) | 8 (8)
Change in visual acuity (Eye disorders) | 23 (23) | 20 (20)
Abnormal blood chemistries (other than liver) (Metabolism and nutrition disorders) | 10 (10) | 13 (13)
Hypoglycemia (Endocrine disorders) | 21 (21) | 9 (9)
Depression (Psychiatric disorders) | 103 (103) | 92 (92)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 55 (55) | 50 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No